CLINICAL TRIAL: NCT07391163
Title: The Possible Protective Role of N-Acetylcysteine Against Oxaliplatin-Induced Peripheral Neuropathy in Patients With Colorectal Cancer
Brief Title: Protective Effect of N-acetylcysteine on Oxaliplatin-Induced Neuropathy in Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Zeyad Khairy Hegazy, Pharmacist & Clinical Researcher, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 36264MS490/1/24
Record Dates: First submitted 2026-01-13; First posted 2026-02-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Oxaliplatin; Peripheral Neuropathy; N-Acetylcysteine; Oxaliplatin Induced Peripheral Neuropathy
MeSH Terms: conditions — Colorectal Neoplasms; Peripheral Nervous System Diseases | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: This is a Randomized, placebo-controlled, parallel-group study. Forty-six patients with stage III colorectal cancer and high-risk stage II will be randomly assigned in a 1:1 ratio to one of two arms:
  Arm 1 (Placebo Group, n=23): Patients will receive 4-6 cycles of modified FOLFOX-6 chemotherapy (Oxaliplatin, Leucovorin, and 5-Fluorouracil) plus oral placebo tablets throughout the chemotherapy cycles.
  Arm 2 (Drug / Experimental Group, n=23): Patients will receive the same chemotherapy regimen in addition to oral N-Acetyl Cysteine 1200 mg administered 1 hour before Oxaliplatin infusion throughout chemotherapy cycles.
  Patients will be recruited from the Oncology Department, Tanta University Hospital, Egypt. Randomization will be done using a sealed envelope method. Standard antiemetic and gastric prophylaxis therapy (IV 5-HT3
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAC Group (Experimental): Patients receive modified FOLFOX-6 chemotherapy plus oral N-acetyl cysteine 1200 mg administered 1 hour before oxaliplatin throughout chemotherapy cycles.
  Interventions: Drug: N-Acetyl Cysteine; Drug: Modified FOLFOX-6 regimen
- Placebo Group (Placebo Comparator): Patients receive modified FOLFOX-6 chemotherapy plus oral placebo tablets administered 1 hour before oxaliplatin throughout chemotherapy cycles.
  Interventions: Drug: Placebo; Drug: Modified FOLFOX-6 regimen

INTERVENTIONS:
Drug: Placebo — Oral placebo tablets identical in appearance to N-acetyl cysteine, administered 1 hour before oxaliplatin throughout chemotherapy cycles.
  Arms: Placebo Group
Drug: N-Acetyl Cysteine — Oral N-acetyl cysteine 1200 mg administered 1 hour before oxaliplatin throughout chemotherapy cycles.
  Arms: NAC Group
Drug: Modified FOLFOX-6 regimen — Oxaliplatin 85 mg/m² IV, leucovorin 400 mg/m² IV, followed by 5-fluorouracil bolus and continuous infusion every 2 weeks.

SUMMARY:
This study investigates the possible protective role of N-Acetylcysteine against oxaliplatin-induced peripheral neuropathy in patients with colorectal cancer. The trial aims to evaluate whether N-Acetylcysteine can reduce the incidence and severity of neuropathy during chemotherapy.

DETAILED DESCRIPTION:
Oxaliplatin, a common chemotherapeutic agent for colorectal cancer, often induces peripheral neuropathy, which can significantly affect patients' quality of life and limit treatment effectiveness. The neuropathy is partly caused by nerve inflammation and oxidative stress.

N-Acetylcysteine (NAC), an antioxidant, has been suggested to protect neurons from oxidative damage and reduce inflammation.

This interventional, randomized, parallel-assignment study will enroll colorectal cancer patients receiving oxaliplatin-based chemotherapy. Participants will be assigned to either receive N-Acetylcysteine alongside chemotherapy or chemotherapy alone. Primary outcomes include the incidence and severity of peripheral neuropathy measured at predefined intervals during treatment.

Secondary outcomes include biochemical markers of nerve inflammation and oxidative stress, including:

* Neurotensin (marker of nerve inflammation)
* Interleukin-6 (marker of systemic inflammation)
* Total Antioxidant Capacity (marker of oxidative stress)

The study aims to provide evidence on whether N-Acetylcysteine can serve as a protective agent against chemotherapy-induced neuropathy, potentially improving treatment tolerance and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged ≥ 18 years old.
* Patients with histologically confirmed diagnosis of Stage III colorectal cancer and high risk Stage II.
* Patients who will be scheduled to receive modified FOLFOX-6.
* Patients with no contraindication to chemotherapy.
* Adequate baseline hematologic values (absolute neutrophilic count ≥ 1.5

  * 109/L, platelet count ≥ 100 × 109/L and hemoglobin level ≥ 10 g/dl).
* Patients with adequate renal function (serum creatinine < 1.5 mg/dl or creatinine clearance (ClCr) ˃ 45 mL/min).
* Patients with adequate liver function (serum bilirubin < 1.5 mg/dl).
* Patients with performance status 0-1 according to Eastern Cooperative Oncology Group (ECOG) score.

Exclusion Criteria:

* Children < 18 years old.
* Prior exposure to chemotherapy.
* Patients with diabetes and other conditions that predispose to neuropathy.
* History of known allergy to oxaliplatin or other platinum agents.
* Concomitant use of any drug has anti-oxidant activity or neuroprotective agent.
* Patients take any medication that increase acetyle choline either central or peripheral.
* Patient was any cardiac disease.
* Pregnant and breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
NCI-CTCAE, Version 5, 2017 | Adverse events will be assessed using NCI-CTCAE v5.0 at baseline (Day 1, prior to Cycle 1) and after Cycle 2 (Day 15) and after Cycle 4 (Day 29). Each chemotherapy cycle lasts 14 days.
  The CTCAE is an international classification system used to assess and describe adverse events resulting from medical treatments, especially in cancer therapy, chemotherapy, and radiation therapy.
  It provides standard criteria to grade the severity of each adverse event on a scale from 1 to 5:
  Grade 1 (Mild): Mild symptoms, no intervention needed.
  Grade 2 (Moderate): Symptoms require minimal intervention or slightly affect daily activities.
  Grade 3 (Severe): Symptoms significantly impact daily activities or require medical intervention.
  Grade 4 (Life-threatening): Life-threatening symptoms requiring urgent intervention.
  Grade 5 (Death): Death due to the adverse event.
FACT/GOG-Ntx-12 | Neurotoxicity-related adverse events will be assessed using the FACT/GOG-Ntx-12 at baseline (Day 1, prior to Cycle 1) and after Cycle 2 (Day 15) and after Cycle 4 (Day 29). Each chemotherapy cycle lasts 14 days.
  The FACT/GOG-Ntx-12 is a patient-reported outcome measure designed to assess chemotherapy-induced neurotoxicity, particularly from drugs such as platinum agents or taxanes.
  It consists of 12 items evaluating peripheral neuropathy symptoms, including numbness, tingling, pain, weakness in hands or feet, and difficulty with walking or handling objects.
  Each item is scored on a 0-4 scale (0 = not at all, 4 = very much), providing a total score reflecting the severity of neurotoxicity.
  It is primarily used to monitor the impact of chemotherapy on neurological function and related quality of life.
BPI-SF | Pain severity and interference will be assessed using the BPI-SF at baseline (Day 1, prior to Cycle 1) and after Cycle 2 (Day 15) and after Cycle 4 (Day 29). Each chemotherapy cycle lasts 14 days.
  The BPI-SF (Brief Pain Inventory - Short Form) is a patient-reported questionnaire used to assess pain severity and its impact on daily functioning.
  It includes questions about the intensity of pain (e.g., worst, least, average, and current pain) and how pain interferes with activities such as walking, work, mood, sleep, and relationships.
  Each item is rated on a 0-10 numeric scale (0 = no pain / no interference, 10 = worst imaginable pain / complete interference), allowing calculation of overall pain severity and interference scores.
  It is widely used in cancer patients and other chronic pain conditions to monitor pain and response to treatment.

SECONDARY OUTCOMES:
Serum IL-6 as a marker of inflammation | IL-6 will be measured at pre-oxaliplatin infusion (baseline) and after infusion completion (post-dose) on Day 1 of Cycle 1 in both study arms. NAC is administered orally 1 hour before baseline sample in the intervention arm. Each FOLFOX cycle is 14 days.
  Serum IL-6 is a pro-inflammatory cytokine commonly used as a biomarker of inflammation.
  Elevated IL-6 levels indicate activation of inflammatory pathways, which can occur due to cancer, chemotherapy, or other physiological stressors.
  Measurement of serum IL-6 allows monitoring of systemic inflammatory responses in patients undergoing chemotherapy.
Serum total anti-oxidant capacity (TAC) as a biomarker of oxidative stress | TAC will be measured at pre-oxaliplatin infusion (baseline) and after infusion completion (post-dose) on Day 1 of Cycle 1 in both study arms. NAC is administered orally 1 hour before baseline sample in the intervention arm. Each FOLFOX cycle is 14 days.
  Serum total antioxidant capacity (TAC) is a biomarker of oxidative stress, reflecting the overall ability of the serum to neutralize free radicals and reactive oxygen species.
  TAC is used to evaluate oxidative damage and antioxidant defense mechanisms, which can be affected by chemotherapy.
Serum neurotensin as a biomarker for neuropathy | NT will be measured at pre-oxaliplatin infusion (baseline) and after infusion completion (post-dose) on Day 1 of Cycle 1 in both study arms. NAC is administered orally 1 hour before baseline sample in the intervention arm. Each FOLFOX cycle is 14 days.
  Description:
  Serum neurotensin (NT) is a peptide biomarker used to assess chemotherapy-induced neuropathy.
  Changes in serum neurotensin levels correlate with peripheral nerve damage and neurotoxic effects caused by chemotherapeutic agents.

CONTACTS AND LOCATIONS:
Overall Officials: Nehal Mohamed Elmashad, Professor, Principal Investigator — Department of Clinical Oncology ,Tanta University School of Medicine
Locations (1):
- Tanta University - Faculty of Medicine ,oncology department, Tanta university hospital., Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. This decision is due to patient privacy and confidentiality concerns, as well as the limited resources available for data sharing in this investigator-initiated study.

REFERENCES:
- [Background] Bazzano G, D'Elia JA, Olson RE. Monosodium glutamate: feeding of large amounts in man and gerbils. Science. 1970 Sep 18;169(3951):1208-9. doi: 10.1126/science.169.3951.1208. PMID 5450696
- [Background] Rome RM. Early diagnosis of gynaecological malignancy. Aust Fam Physician. 1983 Nov;12(11):778-82. PMID 6320789
- [Background] Baidoun F, Elshiwy K, Elkeraie Y, Merjaneh Z, Khoudari G, Sarmini MT, Gad M, Al-Husseini M, Saad A. Colorectal Cancer Epidemiology: Recent Trends and Impact on Outcomes. Curr Drug Targets. 2021;22(9):998-1009. doi: 10.2174/1389450121999201117115717. PMID 33208072
- [Background] Tardiolo G, Bramanti P, Mazzon E. Overview on oxidative stress and inflammation induced by chemotherapy. International Journal of Molecular Sciences. 2019;20(15):3771.